CLINICAL TRIAL: NCT04372745
Title: Evaluation of Home Pregnancy Test by Lay Users Study
Brief Title: Home Pregnancy Test Evaluation, Lay User Study
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-1146
Record Dates: First submitted 2020-04-21; First posted 2020-05-04 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a performance evaluation study to assess the performance of a home pregnancy test (HPT) in the hands of lay users by comparing their results, when used according to the Instructions for Use (IFU), to (a) the lay user confirmed pregnancy status, as determined by a CE marked product, and (b) to trained technicians testing the same urine samples.

The study will also assess the lay user's ability to correctly read results from randomised standards, in addition to leaflet comprehension and product ease of use.

DETAILED DESCRIPTION:
This is an observational study, designed to assess the performance of a home pregnancy test.

The study aims to recruit at total 120 volunteers, being approximately equal numbers of 'pregnant' and not-pregnant' women. Volunteers will be recruited either via direct invitation or advertisement and will attend the study site for one visit lasting 30-40 minutes

Written informed consent will be obtained from all volunteers prior to starting the study.

All volunteers will be issues a unique study number on admission to the study. All data and samples collected will be anonymised throughout the study.

Volunteers will be provided with one investigational home pregnancy test and instructions for use. They will be asked to conduct the test, following the product instructions to obtain a test result which will be recorded on the result sheet. Volunteers will be instructed the product is investigational and the results should not be relied upon to determine their pregnancy status.

Study volunteers will then be interviewed by the study technician, with regards to their understanding of the product instructions and complete an ease of use questionnaire. The comprehension interview may be recorded.

The study technician will then perform 2 further investigational home pregnancy tests on randomised urine standards and the volunteer will read the results.

Finally, the study technician will test the volunteer's urine sample with a marketed pregnancy test and record these results on the results sheet. The results of this test will be used to provide the volunteer with her pregnancy status at the end of the study.

Urine samples provided by the volunteers will be tested with the investigational HPT by an independent technician and also measured for hCG by quantitative immunoassay. Samples may also be measured for other hormones related to pregnancy and fertility.

With participant permission, the samples may be retained frozen within the SPD BioBank and used for future product evaluation or research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Willing to give informed consent
* Willing to conduct a personal home pregnancy test and reveal their pregnancy status
* Seeking to conceive, wishing to conduct a pregnancy test or having recently found out they are pregnant

Exclusion Criteria:

* Currently or previously employed by SPD, Abbott, Alere, Unipath, P&G or affiliates
* Has an immediate relative currently or previously (within last 5 years) employed by SPD, Abbott, Alere, Unipath or P&G, or affiliates
* Healthcare professionals (HCP's) with professional experience either using lateral flow-based devices or conducting near patient testing
* If pregnant, known to be beyond the first trimester (defined as last menstrual period, LMP +13 weeks)
* aken a hormonal preparation containing hCG in the last month, e.g. Pregnyl ®
* Has previously taken part in this study
* Seen the product within the past 6 months

Immediate relatives are defined as parents, children, siblings or partner/spouse

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female only
Study Population: Female volunteers representative of home pregnancy test users.
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Agreement with pregnancy status | 3 months
  The accuracy of the investigational HPT will be calculated against the confirmed pregnancy status of the sample. The corresponding 95% confidence interval will also be calculated for the measure.

SECONDARY OUTCOMES:
Agreement with technician results | 3 months
  The agreement between the lay-user and technician results when both testing the same sample with the investigational HPT as per the IFU. The corresponding 95% confidence interval will also be calculated for the measure.
Comprehension of instructions for use | 3 months
  The percentage number of correct answers in the IFU comprehension exercise
Ease of product use | 3 months
  The cumulative Likert scores for ease of use questions on the device usability questionnaire will be calculated, using a 7 point likert scale, where 1 is equivalent to very easy and 7 is equivalent to very difficult.
Ability to read result | 3 months
  The agreement between the lay-user read of a investigational HPT tested with a spiked standard against the expected result of the spiked standard. The corresponding 95% confidence interval will also be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Principal Investigator — SPD Development Company Ltd
Locations (1):
- SPD Development Company Ltd, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No